CLINICAL TRIAL: NCT04413799
Title: Paravertebral Block Versus Simultaneous Ketamine and Lidocaine Infusions for Pain Management in Rib Fracture Patients
Brief Title: PVB vs Ketamine/Lidocaine in Rib Fracture Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: not enough enrollment
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Susan Kartiko, Assistant Professor of Surgery, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRC1972020
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Rib Fractures; Rib Trauma; Rib Fracture Multiple; Pain, Acute
MeSH Terms: conditions — Rib Fractures; Acute Pain | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- lidocaine/ ketamine infusion (Active Comparator): Lidocaine/ ketamine infusion will be monitored and titrated as necessary by Anesthesiologist led Acute Pain Service.
  Interventions: Combination Product: lidocaine, ketamine intravenous infusion
- paravertebral block with ropivacaine (Active Comparator): Paravertebral block catheter will be placed by Anesthesiology led Acute Pain Service. Once the catheter is inserted, a ropivacaine bolus and infused with ropivacaine, monitored and titrated as necessary by Anesthesiologist led Acute Pain Service.
  Interventions: Drug: paravertebral block with ropivicaine

INTERVENTIONS:
Combination Product: lidocaine, ketamine intravenous infusion — Patients will be started with our standard analgesia regiment which is standing oral acetaminophen 1000mg every 8 hours, ibuprofen 600mg every 6 hours or celecoxib 200mg every 12 hours, and narcotics as needed. All patients who failed the standard analgesia regimen will be approached for the study. Failure of standard analgesia regimen will be determined by respirations >20 minute, tidal volume ≤50% of predicted, numeric pain score ≥ 5, and a poor cough as determined by the trauma team.
  Once the consent is obtained, the patients will be randomized to either PVB (control) or lidocaine/ketamine (study) groups. If the patient is randomized to lidocaine/ketamine group, the anesthesiologist led Acute Pain Service (APS) will prescribe lidocaine/ ketamine infusion, which will be monitored and titrated as necessary by APS. Standard analgesia will be continued on both study groups
  Arms: lidocaine/ ketamine infusion
Drug: paravertebral block with ropivicaine — Patients will be started with our standard analgesia regiment which is standing oral acetaminophen 1000mg every 8 hours, ibuprofen 600mg every 6 hours or celecoxib 200mg every 12 hours, and narcotics as needed. All patients who failed the standard analgesia regimen will be approached for the study. Failure of standard analgesia regimen will be determined by respirations >20 minute, tidal volume ≤50% of predicted, numeric pain score ≥ 5, and a poor cough as determined by the trauma team.
  Once the consent is obtained, the patients will be randomized to either PVB (control) or lidocaine/ketamine (study) groups. If the patient is randomized to PVB, the anesthesiologist led Acute Pain Service (APS) will place a paravertebral block catheter. Ropivacaine infusion will be started, monitored and titrated as necessary by APS. Standard analgesia will be continued on both study groups
  Arms: paravertebral block with ropivacaine

SUMMARY:
Rib fractures are a common admission to the trauma service. The mainstay of treatment is pain control to improve respiratory effort in order to offset the risk of pneumonia and mechanical ventilation. In addition to standard pain control modalities, the investigator's institution utilizes paravertebral blocks as well as lidocaine and ketamine infusions for pain control. The current standard of care for pain control is to begin with acetaminophen, ibuprofen or celecoxib and opioids with the addition of paravertebral blocks as needed. In certain situations, a paravertebral block is contraindicated, and pain control is relegated to lidocaine and ketamine infusion. The use of lidocaine infusion alone and ketamine infusion alone for pain control has been studied and has been shown to be safe. However, concurrent use of these two medications to control rib fracture pain is relatively new and the efficacy compared to paravertebral block is not known. The goal of the study is to show non-inferiority of simultaneous lidocaine and ketamine infusions versus paravertebral blocks.

DETAILED DESCRIPTION:
Traumatic rib fractures are a common pathology in the trauma population. It is estimated that 10% of all trauma patients have rib fractures. The mainstay of treatment of rib fracture is pain control to allow for good pulmonary hygiene and function. When pain is not controlled, patients have a higher chance of developing pneumonia, which can lead to respiratory failure needing mechanical ventilation, eventually increasing patients' morbidity and mortality. These sequelae are most common in the elderly population. Multiple studies has shown that elderly patients with rib fractures have worse outcomes compared to younger patients with the same fracture pattern.

Pain control for acute rib fracture is achieved using multimodal analgesia to reduce the usage of opioids. Multimodal analgesia means using 2 or more drugs that act by different mechanism to provide pain control. The benefit of multimodal strategy is twofold; decrease the use of opioids and the associated side effects (eg. depressed respiratory drive, delirium, alteration of mental status) and better pain control. However, even with multimodal analgesia, pain control for acute traumatic rib fractures can be challenging. There are currently no validated management guidelines for traumatic rib fracture pain control and the approach varies by organization. At the investigator's institution, the investigators use a scheduled regimen of acetaminophen and NSAIDs, along with opioid medication as needed for pain. If this regimen is insufficient, other adjuncts such as paravertebral blocks (PVBs) and intravenous ketamine and lidocaine infusions are utilized. There are currently limited data on the combined use of ketamine and lidocaine infusions for traumatic rib fractures and it is unclear if the combination is non-inferior to PVBs in this patient population.

Continuous PVB infusion is a well-documented approach for pain control in traumatic rib fractures. But, there are occasionally prohibitive situations that contraindicate PVBs, such as vertebral fractures. Ketamine and lidocaine infusions are an attractive alternative in these situations, but the data regarding efficacy are lacking. Low dose ketamine infusion is a new addition to the pain control algorithm for trauma patients. Given that this is a novel approach, studies evaluating efficacy are sparse. There have been two randomized controlled trials utilizing low dose ketamine in trauma patients and elderly patients with rib fractures. Both were unable to show a decrease in opioid use; however, the authors were able to show a decrease in pain scores in patients with injury severity score (ISS) >15 in both studies. Another study of ketamine infusion in traumatic rib fracture patients admitted to the ICU showed an improvement in numeric pain scores (NPS) and decreased opioids requirements but, as in the previous studies, the ISS of these patients was very high (40) in both the ketamine and non-ketamine groups making generalization to the overall trauma population difficult.

Lidocaine has also been extensively studied as a local anesthetic and more recently has become popular as an infusion for systemic pain control. A recent review article compared 16 randomized control trials of lidocaine infusion on postoperative patients and showed that patients undergoing abdominal surgery had significant decreases in postoperative opioid consumption and improved pain scores. There has been some research into lidocaine infusions in burn patients showing that it can decrease opioid usage by 25%, but the cohort was small and there was no difference in reported pain scores. These data are intriguing but the applicability to trauma patients is questionable. Unfortunately, there has been no study to assess lidocaine infusions in patients with traumatic rib fractures. The investigators believe that there is a role for simultaneous lidocaine and ketamine infusions in traumatic rib fracture patients that may provide better pain control than each one used as a single infusion. The investigators propose a prospective, randomized open label clinical trial evaluating continuous infusion of ropivacaine via PVBs against simultaneous ketamine and lidocaine infusions. The instigators hypothesize that simultaneous lidocaine and ketamine infusions is non inferior to PVBs in traumatic rib fracture patients. The results of this study could help guide pain control strategies in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 with rib fracture requiring hospitalization
* Failure of standard pain regimen as determined by RR > 20, TV < or equal to 50% predicted, NPS > or equal to 5, Poor cough

Exclusion Criteria:

* age less than 18 years
* greater than 80 years
* GCS less than or equal to 13
* intubated at admission
* prior or anticipated exploratory laparotomy during this admission
* prior or expected thoracotomy during this admission
* prior or expected emergent craniotomy during this admission
* spinal cord injury
* pelvic injury that has required or will require operative intervention
* inability to accomplish activities of daily living independently
* pregnancy
* incarceration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Score (NPS) | throughout patients' hospitalization time, an average of 1 week
  Numeric pain score is a scale of 1- 10 to ascertain patient's subjective pain severity. Patients will be asked their NPS daily.
Oral Morphine Equivalence (OME) | throughout patients' hospitalization time, an average of 1 week
  Oral morphine equivalence is used to standardized the amount of opioid patient is using regardless the type of opioid that the patient is prescribed.

SECONDARY OUTCOMES:
Hospital Length of Stay (LOS) | captured after patient is discharged, an average of 1 week
  The hospital length of stay will be captured after patient is discharged from the hospital.
ICU Length of Stay (ICU LOS) | captured after patient is discharged, an average of 1 week
  The ICU length of stay will be captured after patient is discharged from the hospital.
incidence of pneumonia | throughout patients' hospitalization time, an average of 1 week
  The diagnosis of pneumonia is captured when it is diagnosed by the primary team taking care of the patient.
ventilator days | throughout patients' hospitalization time, an average of 1 week
  We will obtain the number of days patient is on the ventilator
disposition upon discharge | captured after patient is discharged, an average of 1 week
  Patient's disposition after discharge will be recorded. Disposition of patient will be recorded as home, long term acute facility, skilled nursing facility or acute rehab
in-hospital mortality | captured after patient is discharged, an average of 1 week
  Patient's death will be recorded if it happen before discharge

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Bulger EM, Edwards T, Klotz P, Jurkovich GJ. Epidural analgesia improves outcome after multiple rib fractures. Surgery. 2004 Aug;136(2):426-30. doi: 10.1016/j.surg.2004.05.019. PMID 15300210
- [Background] Bulger EM, Arneson MA, Mock CN, Jurkovich GJ. Rib fractures in the elderly. J Trauma. 2000 Jun;48(6):1040-6; discussion 1046-7. doi: 10.1097/00005373-200006000-00007. PMID 10866248
- [Background] Holcomb JB, McMullin NR, Kozar RA, Lygas MH, Moore FA. Morbidity from rib fractures increases after age 45. J Am Coll Surg. 2003 Apr;196(4):549-55. doi: 10.1016/S1072-7515(02)01894-X. PMID 12691929
- [Background] Karmakar MK, Critchley LA, Ho AM, Gin T, Lee TW, Yim AP. Continuous thoracic paravertebral infusion of bupivacaine for pain management in patients with multiple fractured ribs. Chest. 2003 Feb;123(2):424-31. doi: 10.1378/chest.123.2.424. PMID 12576361
- [Background] Luyet C, Herrmann G, Ross S, Vogt A, Greif R, Moriggl B, Eichenberger U. Ultrasound-guided thoracic paravertebral puncture and placement of catheters in human cadavers: where do catheters go? Br J Anaesth. 2011 Feb;106(2):246-54. doi: 10.1093/bja/aeq309. Epub 2010 Nov 25. PMID 21112880
- [Background] Womack J, Pearson JD, Walker IA, Stephens NM, Goodman BA. Safety, complications and clinical outcome after ultrasound-guided paravertebral catheter insertion for rib fracture analgesia: a single-centre retrospective observational study. Anaesthesia. 2019 May;74(5):594-601. doi: 10.1111/anae.14580. Epub 2019 Jan 27. PMID 30687939
- [Background] Malekpour M, Hashmi A, Dove J, Torres D, Wild J. Analgesic Choice in Management of Rib Fractures: Paravertebral Block or Epidural Analgesia? Anesth Analg. 2017 Jun;124(6):1906-1911. doi: 10.1213/ANE.0000000000002113. PMID 28525509
- [Background] Carver TW, Kugler NW, Juul J, Peppard WJ, Drescher KM, Somberg LB, Szabo A, Yin Z, Paul JS. Ketamine infusion for pain control in adult patients with multiple rib fractures: Results of a randomized control trial. J Trauma Acute Care Surg. 2019 Feb;86(2):181-188. doi: 10.1097/TA.0000000000002103. PMID 30376537
- [Background] Kugler NW, Carver TW, Juul J, Peppard WJ, Boyle K, Drescher KM, Szabo A, Rein L, Somberg LB, Paul JS. Ketamine infusion for pain control in elderly patients with multiple rib fractures: Results of a randomized controlled trial. J Trauma Acute Care Surg. 2019 Nov;87(5):1181-1188. doi: 10.1097/TA.0000000000002479. PMID 31425468
- [Background] Walters MK, Farhat J, Bischoff J, Foss M, Evans C. Ketamine as an Analgesic Adjuvant in Adult Trauma Intensive Care Unit Patients With Rib Fracture. Ann Pharmacother. 2018 Sep;52(9):849-854. doi: 10.1177/1060028018768451. Epub 2018 Apr 2. PMID 29607659
- [Background] de Rocquigny G, Dubecq C, Martinez T, Peffer J, Cauet A, Travers S, Pasquier P. Use of ketamine for prehospital pain control on the battlefield: A systematic review. J Trauma Acute Care Surg. 2020 Jan;88(1):180-185. doi: 10.1097/TA.0000000000002522. PMID 31688832
- [Background] BARTLETT EE, HUTSERANI O. Xylocaine for the relief of postoperative pain. Anesth Analg. 1961 May-Jun;40:296-304. No abstract available. PMID 14448503
- [Background] Kim YC, Castaneda AM, Lee CS, Jin HS, Park KS, Moon JY. Efficacy and Safety of Lidocaine Infusion Treatment for Neuropathic Pain: A Randomized, Double-Blind, and Placebo-Controlled Study. Reg Anesth Pain Med. 2018 May;43(4):415-424. doi: 10.1097/AAP.0000000000000741. PMID 29381569
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Background] Abdelrahman I, Steinvall I, Elmasry M, Sjoberg F. Lidocaine infusion has a 25% opioid-sparing effect on background pain after burns: A prospective, randomised, double-blind, controlled trial. Burns. 2020 Mar;46(2):465-471. doi: 10.1016/j.burns.2019.08.010. Epub 2019 Sep 5. PMID 31493952